CLINICAL TRIAL: NCT00472511
Title: Study of Eyes and Attention Deficit (SEAD)
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Other Study IDs: 2001H0269
Record Dates: First submitted 2007-05-09; First posted 2007-05-11 (Estimated); Last update posted 2008-07-03 (Estimated); Status verified 2008-07

CONDITIONS: ADHD; Convergence Insufficiency; Accommodative Insufficiency
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Ocular Motility Disorders

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Attention-Deficit Hyperactivity Disorder (ADHD) is considered to be one of the most prevalent chronic health conditions in children. It affects between 4% and 12% of young children. A relationship between convergence insufficiency (eye teaming) and ADHD has been shown. However, the effect of ADHD medications on focusing and eye teaming has not been previously investigated. Therefore, the purpose of this study is to determine the effect of ADHD medication on focusing and eye teaming skills.

ELIGIBILITY:
Inclusion Criteria:

* Best corrected visual acuity of 20/25 in both eyes at distance and near;
* Willingness to wear eyeglasses or contact lenses to correct refractive error, if necessary;
* 500" random dot stereopsis

Exclusion Criteria:

* Amblyopia (lazy eye);
* Eye disease

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 75

CONTACTS AND LOCATIONS:
Overall Officials: Levelle Jenkins, OD, Principal Investigator — Ohio State University; Marjean Kulp, OD, MS, Principal Investigator — Ohio State University